CLINICAL TRIAL: NCT03663036
Title: Arthroscopic Superior Capsular Reconstruction With Minimally Invasive Harvested Fascia Lata Autograft - Clinical Outcomes and Survivorship of the Autograft Analysis
Brief Title: Arthroscopic Superior Capsular Reconstruction With Fascia Lata Autograft - Survivorship of the Autograft Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clara Isabel de Campos Azevedo (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Sponsor-Investigator, Clara Isabel de Campos Azevedo, Shoulder Surgery Unit Coordinator, Hospital de Egas Moniz
Organization: Hospital de Egas Moniz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-2018-07HSFX
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Graft Failure; Donor Site Complication; Rotator Cuff Tear
Keywords: Arthroscopic Superior Capsular Reconstruction; Fascia Lata; Autograft; Donor Site Morbidity; Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FL-ASCR (Experimental): Magnetic Resonance Imaging of the shoulder Radiograph of the shoulder
  Interventions: Diagnostic Test: Magnetic Resonance Imaging of the shoulder

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging of the shoulder — Clinical and radiological assessments of the shoulders and the donor sites
  Other Names: Shoulder radiograph; Range of motion and strength measurements

SUMMARY:
An irreparable rotator cuff tear (IRCT) is a challenge, with a controversial definition and different treatment options. None of the latter are exempt of limitations and their survivorship is one of the concerns. In 2013, Mihata et al. proposed a novel treatment option: arthroscopic superior capsular reconstruction using a fascia lata autograft (FL-ASCR) harvested through an open approach. Although no harvest site dysfunction was reported, concerns about donor site morbidity discouraged the use of this type of graft. In 2015, the investigators modified the original FL-ASCR introducing a minimally invasive fascia lata harvesting technique, aiming to reproduce FL-ASCR's promising clinical results in IRCT, while reducing donor site morbidity.

The investigators aim to: 1) Evaluate the mid-term outcomes and donor site morbidity impact of FL-ASCR with minimally invasive harvesting; 2) Analyze the mid-term graft integrity to determine its survivorship 3) Establish clinical and imaging graft integrity correlations to guide the future treatment algorithm.

DETAILED DESCRIPTION:
Task 1 - Prospective evaluation of:

1. The mid-term shoulder outcomes of ASCR with minimally invasive harvested fascia lata autograft The objective of this task is to establish the 3 years postoperative clinical and radiological shoulder outcomes of FL-ASCR with minimally invasive harvesting. The secondary purpose of this task is to test if the FL-ASCR outcomes remain constant after the 2-year evaluation.

   Therefore, the FL-ASCR patients included in this study will have completed the preoperative, 6-month and 2-year postoperative evaluations and will undergo a 3-year postoperative evaluation of:
   1. Bilateral shoulder active range of motion (ROM): elevation, abduction and external rotation (with the arm at the side), measured in degrees with the use of an analogic goniometer; and internal rotation, defined as the highest vertebral body that the patient's thumb can reach, converted afterwards to a scale of 1-5 points: lateral thigh=0; buttock=1; sacrum=2; lumbar=3; 12th thoracic vertebra=4; 7th thoracic vertebra=5.);
   2. Bilateral shoulder strength (supraspinatus, infraspinatus, subscapularis and teres minor) measured in kilograms with the use of a digital dynamometer;
   3. Bilateral functional shoulder scores: the simple shoulder test (SST, 1-12 points), the subjective shoulder value (SSV, 0-100%) and the constant score (CS, 1-100 points).
   4. True anteroposterior shoulder view radiograph of the affected shoulder: the acromiohumeral interval (AHI), considering the distance between the top of the humeral head and the undersurface of the acromion, measured using a software measurement tool (PACS, Agfa HealthCare); the RCT arthritis will be graded according to the Hamada revised radiographic classification.
2. The donor site morbidity impact of FL-ASCR with minimally invasive harvesting The objective of this task is to establish the 3-year donor site morbidity subjective impact of FL-ASCR with minimally invasive harvesting. The secondary aim of this task is to test our hypothesis that the subjective impact of the donor site morbidity after FL-ASCR does not change significantly from the 2-year to the 3-year evaluation. Therefore, at the 3-year evaluation, the patients will be required to answer to the same three closed-ended questions that were asked at the 2-year evaluation to assess the donor site morbidity's impact on the patient's overall satisfaction of the surgical procedure: "Does the harvested thigh bother you?", "Does your shoulder surgery's end result compensate for your thigh's changes?", "Would you undergo the same surgery again?". Accordingly, the patients will also be asked asked, in a closed-ended questionnaire, if they noticed any of the following donor site changes: deformity, pain, numbness and specific donor site-related claudication.

Task 2 - Analysis of the mid-term graft integrity on the 3-year postoperative magnetic resonance imaging (MRI) to determine the graft mid-term survivorship

The objective of this task is to determine the 3-year postoperative survivorship of the graft, establishing the fascia lata superior capsular graft tearing rate and the most frequent site of graft failure at 3 years. A 1.5 Tesla MRI scanner (Siemens Magnetom, U.S.A.) will be used to acquire images in the coronal [proton density fat-saturated (PD FAT-SAT) and T1-weighted], sagittal (PD FAT-SAT and T2 FAT-SAT) and axial (T2* and PD) planes. We and, after blinding, two other independent experienced musculoskeletal radiologists will assess the MRI-images from each patient, in order to:

1. Identify any discontinuity of the graft which, if present, will be classified according to its site as a proximal, an intermediate or a distal tear; and as an anterior or a posterior tear.
2. Identify any discontinuity of the onlay repair of the rotator cuff remnants, which, if present, will be classified a tear of the onlay repair.
3. Grade the supraspinatus, infraspinatus, teres minor and subscapularis muscle fatty degeneration according to the Goutallier et al. classification.
4. Grade the RCT tendon remnants retraction in the coronal plane according to the Patte classification.
5. Grade the supraspinatus muscle atrophy according to the Thomazeau et al. classification.
6. Grade the supraspinatus muscle atrophy according to the tangent sign. The graft survivorship according to the three separate evaluations will be compared to establish the inter-observer reliability of the MRI graft survivorship results.

The type of progression of graft integrity will be determined by comparing the 6-month with the 3-year MRI evaluation of the graft survivorship.

Task 3 - Comparative analysis of the clinical, radiological and MRI preoperative and postoperative variables

The objective of this task is to find correlations between the graft survivorship and the results from tasks 1 and 2. The aim is to establish the clinical importance of mid-term graft survivorship.

The investigators will compare the ROM, shoulder strength, SSV, SST, CS and AHI from preoperative to 3 years postoperative; and from 2 years postoperative to 3 years postoperative (paired-samples t-test). The investigators will compare all continuous variables between the group of ASCR patients who underwent an additional onlay partial RCT repair and the group that underwent ASCR without an onlay partial RCT repair, between the anterior acromioplasty-ASCR group and the group that did not undergo an anterior acromioplasty, between the tenotomy-ASCR group and the no-LHBT group, between the preoperative and postoperative AHI<7mm group and the AHI≥7mm group, and between the intact-graft group and the graft-tear group (Mann-Whitney U test). The investigators will compare all categorical variables, including the donor site morbidity and overall subjective outcome results, between the groups (Fisher's exact test).

To determine the repercussion of FL-ASCR and of the graft integrity on the rotator cuff muscle function the investigators will compare the progression of the Goutallier classification of each rotator cuff muscle from preoperative to 3 years postoperative, as well as the cumulative Goutallier score (the sum of the fatty infiltration stages of the four muscles) and the global fatty muscle degeneration index (the mean value of the grades for the supraspinatus, infraspinatus, and subscapularis), between the intact-graft group and the graft-tear group.

A significant difference will be defined as P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* FL-ASCR by the same surgeon (principal investigator) since 2015
* completed the preoperative and the 6 months postoperative clinical, radiological and MRI assessments

Exclusion Criteria:

* secondary surgery for the removal of the implanted autograft in the shoulder which had previously ungergone the FL-ASCR procedure
* secondary surgery to the harvested thigh

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Shoulder outcomes of FL-ASCR with minimally invasive harvesting at 3 years postoperative | 2 years
  Bilateral shoulder active range of motion (ROM): elevation (0 -180º), abduction (0 -180º) and external rotation (0 -100º), measured in degrees ; and internal rotation, defined as the highest vertebral body that the patient's thumb can reach, converted afterwards to a scale of 1-5 points: lateral thigh=0; buttock=1; sacrum=2; lumbar=3; 12th thoracic vertebra=4; 7th thoracic vertebra=5.). Bilateral functional shoulder scores: the simple shoulder test (SST, 1-12 points), the subjective shoulder value (SSV, 0-100%) and the constant score (CS, 1-100 points). Bilateral shoulder strength (supraspinatus, infraspinatus, subscapularis and teres minor, 0 -15 kg). For every scale range provided, higher values represent a better outcome.

SECONDARY OUTCOMES:
Autograft mid-term survivorship at 3 years postoperative | 2 years
  Analysis of the mid-term graft integrity on the 3-year postoperative magnetic resonance imaging (scale: 0 -1): 0 = graft absent or not healed to the greater tuberosity/superior glenoid; 1 = graft present and healed to the greater tuberosity and superior glenoid. For the scale range provided, higher values represent a better outcome.
Fascia lata minimally invasive harvesting donor site morbidity impact at 3 years postoperative | 2 years
  Three closed-ended questions to assess the donor site morbidity's impact on the patient's overall satisfaction of the surgical procedure will be asked to the participants: "Does the harvested thigh bother you?" (scale: , "Does your shoulder surgery's end result compensate for your thigh's changes?" (scale: 0 - 1; 0 = no, 1 = yes), "Would you undergo the same surgery again?" (scale: 0 - 1; 0 = no, 1 = yes). The participants will be asked, in a closed-ended questionnaire, if they noticed any of the following donor site changes: deformity (scale: 0 - 1; 0 = no, 1 = yes), pain (scale: 0 -1; 0 = no, 1 = yes), numbness (scale: 0 - 1; 0 = no, 1 = yes)and specific donor site-related claudication (scale: 0 -1; 0 = no, 1 = yes). For every scale range provided, higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clara IC Azevedo, MD, Principal Investigator — Centro Hospitalar de Lisboa Ocidental
Locations (1):
- Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Campos Azevedo CI, Angelo ACLPG, Vinga S. Arthroscopic Superior Capsular Reconstruction With a Minimally Invasive Harvested Fascia Lata Autograft Produces Good Clinical Results. Orthop J Sports Med. 2018 Nov 27;6(11):2325967118808242. doi: 10.1177/2325967118808242. eCollection 2018 Nov. PMID 30505873
- [Background] Angelo ACLPG, de Campos Azevedo CI. Minimally invasive fascia lata harvesting in ASCR does not produce significant donor site morbidity. Knee Surg Sports Traumatol Arthrosc. 2019 Jan;27(1):245-250. doi: 10.1007/s00167-018-5085-1. Epub 2018 Aug 1. PMID 30069653
- [Derived] Azevedo CIC, Catarina Leiria Pires Gago Angelo A, Campos-Correia D, Delgado L, Ferreira N, Sevivas N. Clinical Importance of Graft Integrity in Arthroscopic Superior Capsular Reconstruction Using a Minimally Invasively Harvested Midthigh Fascia Lata Autograft: 3-Year Clinical and Magnetic Resonance Imaging Outcomes. Am J Sports Med. 2020 Jul;48(9):2115-2128. doi: 10.1177/0363546520928649. PMID 32667265